CLINICAL TRIAL: NCT00283153
Title: Controlled Study of Affect Recognition Training for Individuals With Acquired Brain Injury
Brief Title: Affect Recognition: Enhancing Performance of Persons With Acquired Brain Injury (ABI)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); Massey University (Other); Wake Forest University Health Sciences (Other); Brock University (Other)
Responsible Party: Principal Investigator, Barry Willer, Professor, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DR-050573-BW-2300; NIDRR H133G080043A
Record Dates: First submitted 2006-01-24; First posted 2006-01-27 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: Traumatic Brain Injury; Stroke; Emotion Recognition; Affect; Interventions
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAR (Experimental): Facial affect recognition training (with computer assistance)
  Interventions: Behavioral: Facial Affect Recognition Training
- SEI (Experimental): Stories of Emotional Inference
  Interventions: Other: Stories of Emotional Inference

INTERVENTIONS:
Behavioral: Facial Affect Recognition Training — A series of pictures of faces displaying various emotions are presented one at a time using a computerized training program.Participants are taught to recognize how emotions affect facial features such as the mouth and eyes.Participants are also taught how to recognize their own emotions.
  Arms: FAR
Other: Stories of Emotional Inference — Participants are presented with a series of short stories one at a time. Each story presents various contextual cues regarding the emotions the characters are likely to experience. Participants learn to connect the cues to specific emotions.
  Other Names: Cognitive intervention
  Arms: SEI

SUMMARY:
The purpose of this research is to evaluate the effectiveness of three training programs designed to teach persons with acquired brain injury (ABI) to recognize emotions. It is hypothesized that the training programs will enhance several aspects of emotion recognition in persons with ABI. Furthermore, it is expected that these effects will be maintained over time, and will positively influence participants' social behavior and integration.

DETAILED DESCRIPTION:
Research has demonstrated that persons with acquired brain injury (ABI) often have difficulty recognizing emotions. This includes emotions portrayed in facial expressions, as well as inferring emotions based on social context. The ability to identify emotions in others is an essential component for the engagement of successful social interactions. It has been suggested that a decreased ability to recognize emotions may result in inappropriate behaviors and have a detrimental impact on social relationships. Despite the significance of this problem, very few studies have addressed this need in the ABI population.

Comparisons: Three groups receiving computer-based training programs. Two of the groups are trained to learn how to identify emotions of happy, sad, angry and fearful. The third training experience presents participants with a variety of learning tasks from managing money to grocery shopping.

1. Facial Affect Recognition (FAR) group: This group is shown faces on the computer and asked to identify the emotion being expressed. Subjects are also asked to describe situations that they associate with the emotions being trained, as well as mimic facial expressions in a mirror.
2. Stories of Emotional Inference (SEI) group: This group is asked to read stories on the computer that describe the interaction of events with characters' beliefs, wants and behaviors. From this information, subjects are asked to infer the emotions of the characters throughout the stories.
3. Cognitive Training Group (CTG): This group is given educational experiences in a variety of life skill areas including banking and applying for a job. This training is aimed at resolving some of the frustrations experienced by persons with ABI. Subjects may learn various computer skills including, Word, Excel, Internet Search or Games.

Before and after training, emotion recognition will be measured with pictures of faces; vocal recordings; stories that give the contextual cues to emotion; and hypothetical situations. In addition, participants' cognitive skills, social behavior and integration will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age between eighteen and sixty-five years old.
* At minimum, one year post-injury.
* Glasgow Coma Score (GCS) of 12 or less, or stroke with hemi-paresis signifying a moderate to severe acquired brain injury.
* A TBI that resulted in either a closed or open head injury or a stroke that resulted in severe disability
* Perform at least one standard deviation below the norm on the DANVA2-Adult Faces test, a standardized assessment of facial affect recognition.
* Verbally able to express a basic understanding of emotional descriptors (e.g. Happy, sad, angry, fearful).
* Demonstrate basic comprehension for short paragraphs presented in 2 ways: 1)auditorily and 2)silent reading. This measure is part of the Discourse Comprehension Test.

Exclusion Criteria:

* Diagnosed mental illness.
* Uncorrected visual acuity.
* Uncorrected hearing impairment.
* Perceptual impairment (visual neglect and/or visual discrimination).
* Impaired verbal expression/ aphasia
* Alcohol or substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-10; Primary Completion 2012-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic Assessment of Nonverbal Affect-Adult Faces (DANVA2-AF) | Seven months
Emotional Inference From Stories Test | Seven months

SECONDARY OUTCOMES:
Interpersonal Reactivity Index | Seven Months
Neuropsychiatric Inventory | Seven Months

CONTACTS AND LOCATIONS:
Overall Officials: Barry Willer, Ph.D., Principal Investigator — University at Buffalo, Department of Psychiatry
Locations (4):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - Carolinas HealthCare System, Charlotte, North Carolina
- Brock University, St. Catharines, Ontario, Canada
- Massey University, Wellington, New Zealand

REFERENCES:
- [Background] Zupan B, Neumann D, Babbage DR, Willer B. The importance of vocal affect to bimodal processing of emotion: implications for individuals with traumatic brain injury. J Commun Disord. 2009 Jan-Feb;42(1):1-17. doi: 10.1016/j.jcomdis.2008.06.001. Epub 2008 Jul 9. PMID 18692197
- [Background] Radice-Neumann D, Zupan B, Babbage DR, Willer B. Overview of impaired facial affect recognition in persons with traumatic brain injury. Brain Inj. 2007 Jul;21(8):807-16. doi: 10.1080/02699050701504281. PMID 17676438
- [Background] Radice-Neumann D, Zupan B, Tomita M, Willer B. Training emotional processing in persons with brain injury. J Head Trauma Rehabil. 2009 Sep-Oct;24(5):313-23. doi: 10.1097/HTR.0b013e3181b09160. PMID 19858965
- [Background] Babbage DR, Yim J, Zupan B, Neumann D, Tomita MR, Willer B. Meta-analysis of facial affect recognition difficulties after traumatic brain injury. Neuropsychology. 2011 May;25(3):277-285. doi: 10.1037/a0021908. PMID 21463043
- [Result] Neumann D, Babbage DR, Zupan B, Willer B. A randomized controlled trial of emotion recognition training after traumatic brain injury. J Head Trauma Rehabil. 2015 May-Jun;30(3):E12-23. doi: 10.1097/HTR.0000000000000054. PMID 24842590
- [Result] Zupan B, Babbage D, Neumann D, Willer B. Recognition of facial and vocal affect following traumatic brain injury. Brain Inj. 2014;28(8):1087-95. doi: 10.3109/02699052.2014.901560. Epub 2014 Apr 4. PMID 24701988
- [Result] Yim J, Babbage DR, Zupan B, Neumann D, Willer B. The relationship between facial affect recognition and cognitive functioning after traumatic brain injury. Brain Inj. 2013;27(10):1155-61. doi: 10.3109/02699052.2013.804203. Epub 2013 Jul 29. PMID 23895556
- [Result] Neumann D, Zupan B, Babbage DR, Radnovich AJ, Tomita M, Hammond F, Willer B. Affect recognition, empathy, and dysosmia after traumatic brain injury. Arch Phys Med Rehabil. 2012 Aug;93(8):1414-20. doi: 10.1016/j.apmr.2012.03.009. Epub 2012 Mar 23. PMID 22446155